CLINICAL TRIAL: NCT03890432
Title: GLUCOSAFE 2 - A New Tool for Nutritional Management and Insulin-therapy in the Intensive Care Unit (ICU): Randomized Controlled Study
Brief Title: GLUCOSAFE 2 - A New Tool for Nutritional Management and Insulin-therapy in the Intensive Care Unit (ICU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HEIDEGGER CP (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor-Investigator, HEIDEGGER CP, Privat-Docent, Senior Lecturer, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G2-0219
Record Dates: First submitted 2019-02-14; First posted 2019-03-26 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Energy Supply; Deficiency, Severe; Protein Deficiency; Hypoglycemia; Hyperglycemia
Keywords: Nutrition management; Glycaemia control; ICU; Software; Critical illness; Insulin-therapy; Critically ill patients; Blood glucose control
MeSH Terms: conditions — Critical Illness; Protein Deficiency; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GLUCOSAFE 2 (Experimental): Insulin-therapy and nutrition support guided by the GLUCOSAFE 2 software.
  Interventions: Device: GLUCOSAFE 2
- Local protocol control group (Active Comparator): Insulin-therapy and nutrition support guided by the local protocols (electronic or paper version) of the ICU/HUG.
  Interventions: Device: Local protocol control group with routine care
- Historical control group (Other): Retrospective data with standard care before the beginning of the pilot study in order to minimize the "cross-over" effect due to the fact that caregivers are going to have in charge patients in both groups (intervention and control group) at the same time.
  Interventions: Device: Historical control group with routine care

INTERVENTIONS:
Device: GLUCOSAFE 2 — Use of GLUCOSAFE 2 software for nutrition management and insulin-therapy
  Arms: GLUCOSAFE 2
Device: Local protocol control group with routine care — Use of the local protocols (electronic or paper version) for nutrition management and blood glucose control.
  Arms: Local protocol control group
Device: Historical control group with routine care — Use of the local protocols (electronic or paper version) for nutrition management and blood glucose control.
  Arms: Historical control group

SUMMARY:
The survival and the outcomes of critically ill patients are strongly influenced by insulin-therapy and nutritional support. The GLUCOSAFE 2 pilot study, aims to test the performance and the security of the new GLUCOSAFE 2 software, developed by the model-based medical decision support of Aalborg University (Denmark) and adapted to the clinical needs in the intensive care unit (ICU) of the Geneva University Hospital (HUG). This new device is based on a mathematical model of the glucose-insulin metabolism and attempts to give advices for better glycaemia control and nutritional therapy. The GLUCOSAFE 2 study hypothesizes that the use of the Glucosafe 2 software will allow better glycaemia ("Time-in-target") control and better achievement of nutritional energy and protein targets in comparison to the local protocols.

ELIGIBILITY:
Inclusion Criteria:

All patients ≥ 18 years admitted to the ICU with

* An expected length of stay ≥ 72h
* At least 1 blood glucose (BG) measurement ≥10 mmol/l or 2 BG measurement ≥ 8.5 mmol/l
* Informed Consent signed by the subject/ legal representative, except for patients in the historical control group

Exclusion Criteria:

* Lack of legal consent or consent withdrawn, except for patients in the historical control group
* Pregnant or breast feeding
* Diabetic ketoacidosis or hyperosmolar state
* Oral feeding
* Fulminant hepatic failure
* Medically contraindicated to receive rapidly acting insulin by intravenous (iv) infusion or iv injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Time-in-target (range: 5.0 - 8.5 mmol/l) | During ICU stay, up to 15 days post-randomization.
  Time spent in the glycaemia range of 5.0 - 8.5 mmol/l per day, per patient and in the cohort

SECONDARY OUTCOMES:
Overall number of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events | During ICU stay, up to 15 days post-randomization.
  Overall number of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events (per patient and in the cohort)
Overall percentage of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events | During ICU stay, up to 15 days post-randomization.
  Overall percentage of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events (per patient and in the cohort)
Number of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events due to non-compliance | During ICU stay, up to 15 days post-randomization.
  Overall number of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events due to non-compliance (only in intervention arm)
Percentage of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events due to non-compliance | During ICU stay, up to 15 days post-randomization.
  Percentage of mild (<3.3 mmol/l) and severe (<2.2 mmol/l) hypoglycemia events due to non-compliance (only in intervention arm)
Time to normalize blood glucose (5.0-8.5 mmol/l) | During ICU stay, up to 15 days post-randomization.
  Three values < 8.5 mmol/l as indicator for normalization
Percentage of time in the ICU (per patient and in the cohort) with hyperglycaemia (BG > 8.5 mmol/l) | During ICU stay, up to 15 days post-randomization.
  Percentage of time with BG > 8.5 mmol/l before and after normalization per patient and in the cohort.
Percentage of time in the ICU (per patient and in the cohort) with hyperglycaemia (BG > 8.5 mmol/l) due to non compliance | During ICU stay, up to 15 days post-randomization.
  Percentage of time with BG > 8.5 mmol/l before and after normalization per patient and in the cohort due to non compliance (only in the intervention arm).
Number of hyperglycemic episodes after normalization (> 8.5 mmol/l) | From normalization time during ICU stay, up to 15 days post-randomization.
  Three values < 8.5 mmol/h as indicator for normalization
Number of hyperglycemic episodes after normalization (> 8.5 mmol/l) due to non compliance | From normalization time during ICU stay, up to 15 days post-randomization.
  Three values < 8.5 mmol/h as indicator for normalization
Number of episodes (per patient and in the cohort) where a BG measurements is not followed up within 30 minutes by a request for Glucosafe 2 advice | During ICU stay, up to 15 days post-randomization.
  Number of episodes (per patient and in the cohort) where a BG measurements is not followed up within 30 minutes by a request for Glucosafe 2 advice
Number of episodes (per patient and in the cohort) where pumps were not set within 30 min according to Glucosafe2 advice accepted by the nurse. | During ICU stay, up to 15 days post-randomization.
  Number of episodes (per patient and in the cohort) when pumps were not set within 30 min according to Glucosafe2 advice accepted by the nurse.
Number of advices given by GS2 which were accepted, accepted with modification, or rejected. | During ICU stay, up to 15 days post-randomization.
  Number of advices given by GS2 which were accepted, accepted with modification, or rejected.
Frequency of daily and cumulated BG measurements per patient and in the cohort | During ICU stay, up to 15 days post-randomization.
  Frequency of BG measurements (per patient and in the cohort)
Frequency of daily and cumulated adjustments of insulin and nutrition pump settings (per patient and in the cohort) | During ICU stay, up to 15 days post-randomization.
  Frequency of daily and cumulated adjustments of insulin and nutrition pump settings (per patient and in the cohort)
Glycaemic variability | During ICU stay, up to 15 days post-randomization.
  Mean and standard deviation (SD) of blood glucose measurements. Daily maximum blood glucose difference.
Protein goal achievements (80-100% of accumulated target) with a target of 1.3 g/kg of body weight per day. | During ICU stay, up to 15 days post-randomization.
  Percentage of proteins received per day and at the end of the ICU stay with a target of 1.3 g/kg of body weight per day.
Caloric goal achievements (80-100% of the accumulated target) by indirect calorimetry (IC) or predictive formula if IC not feasible. | During ICU stay, up to 15 days post-randomization.
  Percentage of nutritional and non-nutritional calories received per day and at the end of the ICU stay with a target defined by IC or predictive formula if IC not feasible.
Energy debt: difference between the defined energy target (80-100%, defined by IC or predictive formula) and the energy received (nutritional and non-nutritional) | During ICU stay, up to 15 days post-randomization.
  Per day and at the end of the ICU stay.
Protein debt: difference between the defined protein target (1.3 g/kg of body weight/day) and the proteins received | During ICU stay, up to 15 days post-randomization.
  Per day and at the end of the ICU stay.
Prediction of BG | During ICU stay, up to 15 days post-randomization.
  Prediction error as a function of time elapsed since last BG measurement, per patient, per cohort.measurement (per patient and per cohort).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia P. Heidegger, MD, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Hôpitaux Universitaire de Genève, Geneva, Canton of Geneva
  - Service of Intensive Care, Geneva University Hospital,, Geneva, Canton of Geneva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Watteville A, Pielmeier U, Di Marco M, Gayet-Ageron A, Siegenthaler N, Parel N, Wozniak H, Primmaz S, Pugin J, Andreassen S, Heidegger CP. Glucosafe 2-A new tool for nutritional management and insulin-therapy in the intensive care unit: Randomized controlled study (the Glucosafe 2 protocol). PLoS One. 2025 Mar 4;20(3):e0316624. doi: 10.1371/journal.pone.0316624. eCollection 2025. PMID 40036206